CLINICAL TRIAL: NCT05716100
Title: A Randomized, Double-blind, Placebo-Controlled, Multicenter Phase 3 Study to Evaluate the Safety, Tolerability, and Efficacy of XEN1101 as Adjunctive Therapy in Focal-Onset Seizures
Brief Title: A Randomized Study of XEN1101 Versus Placebo in Focal-Onset Seizures (X-TOLE3)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPF-010-302; 2022-502281-25-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-26; First posted 2023-02-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Focal Onset Seizures
Keywords: Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- XEN1101 25 mg/day (Experimental): XEN1101 25 mg/day
  Interventions: Drug: XEN1101
- XEN1101 15 mg/day (Experimental): XEN1101 15 mg/day
  Interventions: Drug: XEN1101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN1101 — XEN1101 Capsules
  Other Names: Azetukalner
  Arms: XEN1101 15 mg/day; XEN1101 25 mg/day
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
The X-TOLE3 Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study that will evaluate the clinical efficacy, safety and tolerability of XEN1101 administered as adjunctive therapy in focal-onset seizures.

DETAILED DESCRIPTION:
Approximately 360 subjects will be randomized in a blinded manner to one of two active treatment groups or placebo in a 1:1:1 fashion (XEN1101 25 mg : 15 mg : Placebo). Eligible subjects will have up to 9.5 weeks of baseline to assess frequency of seizures, followed by 12 weeks of blinded treatment. In order to be included in the study, subjects must be treated with a stable dose of 1 to 3 allowable antiseizure medications (ASMs) for at least one month prior to screening, during baseline, and throughout the double-blind treatment period (DBP) of the study. During the DBP, subjects will be instructed to orally take XEN1101 or placebo once daily with an evening meal.

Subjects who complete the 12-week DBP will have the opportunity to qualify and enroll in a separate open-label extension (OLE) study for continued treatment with XEN1101. Subjects who do not enroll in the OLE will enter a 8-week post treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study
* Diagnosis (≥2 years) of focal epilepsy according to the International League Against Epilepsy (ILAE) Classification of Epilepsy (2017). Subject must have had adequate trials of at least 2 ASMs, which were given (and tolerated) at adequate therapeutic doses, without achieving sustained seizure freedom.
* Treatment with a stable dose of 1 to 3 allowable current ASMs for at least one month prior to screening, during baseline, and throughout the duration of the DBP
* Able to keep accurate seizure diaries

Exclusion Criteria:

* Previously documented electroencephalogram which shows any pattern not consistent with focal etiology of seizures.
* History of focal aware non-motor seizures only, non-epileptic psychogenic seizure, primary generalized seizure, developmental and epileptic encephalopathy, including Lennox-Gastaut syndrome.
* Seizures secondary to drug or alcohol use, ongoing infection, neoplasia, demyelinating disease, degenerative neurological disease, metabolic illness, progressive structural lesion, encephalopathy, or progressive central nervous system (CNS) disease.
* History of status epilepticus or repetitive seizures within the 12-month period preceding Visit 1 where the individual seizures cannot be counted.
* History of neurosurgery for seizures <1 year prior to Visit 1, or radiosurgery <2 years prior to enrollment.
* Any medical condition or personal circumstance that, in the opinion of the investigator, exposes the subject to unacceptable risk by participating in the study or prevents adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Median percent change (MPC) in focal seizure frequency from baseline to DBP for XEN1101 versus placebo. | From baseline through to the double blind period (week 12).

SECONDARY OUTCOMES:
Proportion of subjects experiencing ≥50% reduction in focal seizure frequency from baseline through the DBP for XEN1101 versus placebo. | From baseline through to the double blind period (week 12).
MPC in weekly (7 days) focal seizure frequency from baseline to Week 1 for XEN1101 versus placebo. | From baseline through to the week 1.
Proportion of subjects experiencing "at least much improved" (including "much" and "very much improved") in Patient Global Impression of Change (PGI-C). | From baseline through to the double blind period (week 12).
To assess adverse events as criteria for safety and tolerability of XEN1101. | From screening through to 56 days post-final dose

CONTACTS AND LOCATIONS:
Overall Officials: Xenon Medical Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (89):
- United States (17):
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Rancho Research Institute, Downey, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California Irvine Health, Orange, California
  - Panhandle Research and Medical Clinic, Gulf Breeze, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - 9D University Health Center, Detroit, Michigan
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Five Towns Neuroscience Research, Woodmere, New York
  - Duke University Clinic, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
- Argentina (12):
  - Hospital Ramos Mejia, Buenos Aires
  - Hospital De Alta Complejidad en Red el Cruce, Buenos Aires
  - Policlinico Lomas, Buenos Aires
  - Instituto de Neurologia Cognitiva (INECO), Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - STAT Resarch S.A., Buenos Aires
  - CENyR Centro de Especialidades Neurologicas y Rehabilitacion, C.a.b.a.
  - FLENI, C.a.b.a.
  - Hospital Córdoba, Córdoba
  - Hospital Central Ramon Carrilo, San Luis
  - Sanatori del Sur S.A., San Miguel de Tucumán
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Alfred Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne
- Austria (3):
  - University Hospital Innsbruck, Innsbruck
  - Universitätsklinik für Neurologie, Salzburg
  - Medical University of Vienna, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Bulgaria (2):
  - MHATNPsy Sveti Naum EAD, Sofia
  - Medical center OPHTHA-NEURO, Sofia
- Chile (4):
  - Clinica Universidad de Los Andes, Santiago
  - Centro de Investigacion Clinica UC, Santiago
  - CINSAN, Santiago
  - Hospital Clínico Viña del Mar, Viña del Mar
- Croatia (5):
  - University Hospital Center Osijek, Osijek
  - Clinical Hospital Center Rijeka, Klinika za Neurologiju, Rijeka
  - Poliklinika Bonifarm, Zagreb
  - University Hospital Center Zagreb, Zagreb
  - Poliklinika LF MEDICAL, Zagreb
- Czechia (3):
  - EUC Hradec Kralove Clinic, Hradec Králové
  - Nemocnicni lekarna FN Motol / Motol University Hospital, Prague
  - Forbeli s.r.o., Prague
- Kuopio University Hospital, Kuopio, Finland
- France (6):
  - Hopital Neurologique Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire de Lille (CHU de Lille), Lille
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Fondation A. de Rothschild, Paris
  - Chu de Rennes Hôpital Pontchaillou, Rennes
  - Hôpital de Hautepierre, Strasbourg
- Germany (3):
  - Universitätsklinikum Aachen, Aachen
  - Krankenhaus Mara gGmbH, Bielefeld
  - University Hospital Frankfurt, ZNN - Epilepsy Center Frankfurt Rhine-Main, Frankfurt
- Semmelweis Egyetem, Idegsebészeti és Neurointervenciós Klinika, Budapest, Hungary
- Israel (4):
  - Hadassah Medical Center, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Ospedali Riuniti di Ancona, Ancona
  - Università degli studi di Bari Aldo Moro, Bari
- Mexico (4):
  - Grupo Medico Camino, Benito Juárez
  - Human Science Research Trials, Mexico City
  - Axis Heilsa S. de R.L. de C.V. Althian, Monterrey
  - Neurocencias Esudios Clinicos S.C., Sinaloa
- Kempenhaeghe, Heeze, Netherlands
- Poland (4):
  - COPERNICUS Podmiot Leczniczy, Gdansk
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Portugal (8):
  - Centro Hospitalar Universitário de Coimbra - CHUC, Coimbra
  - Hospital da Senhora da Oliveira, Guimarães
  - Centro Hospitalar de Lisboa Norte, Lisbon
  - Centro Hospitalar Lisboa Ocidental, Lisbon
  - Centro Hospitalar Universitário de Santo António, Porto
  - Hospital Pedro Hispano, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, Santa Maria da Feira
  - ULS de Trás-os-Montes e Alto Douro, Vila Real
- Spain (3):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Unversitario Ramon y Cajal, Madrid
  - Hospital universitario Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: No